CLINICAL TRIAL: NCT00051558
Title: Comparison of the Effects of Teriparatide With Those of Alendronate Sodium on Lumbar Spine Bone Mineral Density in Glucocorticoid-Induced Osteoporosis
Brief Title: Comparison of Teriparatide With Alendronate for Treating Glucocorticoid-Induced Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6484; B3D-US-GHBZ
Record Dates: First submitted 2003-01-13; First posted 2003-01-14 (Estimated); Results first posted 2009-02-13 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide; Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Teriparatide 20 micrograms/day injection plus oral placebo, 36 months
  Interventions: Drug: Teriparatide; Drug: Placebo
- B (Active Comparator): Alendronate 10 mg/day oral plus injection placebo, 36 months
  Interventions: Drug: Alendronate Sodium; Drug: Placebo

INTERVENTIONS:
Drug: Teriparatide — 20 micrograms/day, injection, 36 months
  Other Names: LY333334; Forteo; Forsteo
  Arms: A
Drug: Alendronate Sodium — 10 mg/day, oral, 36 months
  Arms: B
Drug: Placebo — Oral placebo, daily, 36 months
  Arms: A
Drug: Placebo — Injection placebo, daily, 36 months
  Arms: B

SUMMARY:
Osteoporosis is a condition in which the amount of bone is reduced, the bones are weak, and there is an increased risk for fractures. Glucocorticoids (such as prednisone) are prescribed to treat a large number of conditions such as arthritis and asthma. When taken for several months or longer, glucocorticoids can cause bone loss and lead to a form of osteoporosis called "glucocorticoid-induced osteoporosis." This study compared the effects of teriparatide, the study drug, with alendronate, an approved drug for treating glucocorticoid-induced osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age 21 years or older
* Taking on average 5.0 mg/day prednisone or equivalent for at least 3 months prior to screening

Exclusion Criteria:

* Taking bisphosphonates within past 6 months
* More than 30 micrograms/day of estradiol or equivalent in past 3 months
* History of alcoholism or drug abuse in past year
* Pregnant women or nursing mothers

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2002-11; Primary Completion 2006-07 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- United States (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Loma Linda, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Palo Alto, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Jamestown, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Milwaukee, Wisconsin
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Vienna
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Leuven
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Aarhus, Denmark
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Oslo, Norway
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ponce

REFERENCES:
- [Derived] Saag KG, Agnusdei D, Hans D, Kohlmeier LA, Krohn KD, Leib ES, MacLaughlin EJ, Alam J, Simonelli C, Taylor KA, Marcus R. Trabecular Bone Score in Patients With Chronic Glucocorticoid Therapy-Induced Osteoporosis Treated With Alendronate or Teriparatide. Arthritis Rheumatol. 2016 Sep;68(9):2122-8. doi: 10.1002/art.39726. PMID 27111239
- [Derived] Devogelaer JP, Adler RA, Recknor C, See K, Warner MR, Wong M, Krohn K. Baseline glucocorticoid dose and bone mineral density response with teriparatide or alendronate therapy in patients with glucocorticoid-induced osteoporosis. J Rheumatol. 2010 Jan;37(1):141-8. doi: 10.3899/jrheum.090411. Epub 2009 Nov 16. PMID 19918047
- [Derived] Saag KG, Shane E, Boonen S, Marin F, Donley DW, Taylor KA, Dalsky GP, Marcus R. Teriparatide or alendronate in glucocorticoid-induced osteoporosis. N Engl J Med. 2007 Nov 15;357(20):2028-39. doi: 10.1056/NEJMoa071408. PMID 18003959
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Teriparatide: Teriparatide 20 micrograms/day injection plus oral placebo, 36 months
- Alendronate: Alendronate 10 mg/day oral plus injection placebo, 36 months
Period: Overall Study
Arm/Group | Teriparatide | Alendronate
Started | 214 | 214
Completed | 123 | 118
Not Completed | 91 | 96
Not completed — Adverse Event | 30 | 18
Not completed — Withdrawal by Subject | 29 | 42
Not completed — Death | 9 | 15
Not completed — Lost to Follow-up | 4 | 13
Not completed — Protocol Violation | 3 | 4
Not completed — Protocol Entry Criteria Unmet | 1 | 2
Not completed — Sponsor Decision | 6 | 1
Not completed — Other | 2 | 1
Not completed — Significant Lab Value | 2 | 0
Not completed — Physician Decision | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Alendronate | Total
Number analyzed (Participants) | 214 | 214 | 428
Age, Customized [Number; unit: participants]
  Age < 35 years | 13 | 19 | 32
  35 <= Age < 50 years | 55 | 35 | 90
  50 <= Age < 65 years | 86 | 93 | 179
  Age >= 65 years | 60 (1.518) | 67 (1.528) | 127
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 173 | 345
  Male | 42 | 41 | 83
Region of Enrollment [Number; unit: participants]
  United States | 62 | 64 | 126
  Belgium | 8 | 8 | 16
  Denmark | 4 | 3 | 7
  Austria | 1 | 2 | 3
  Norway | 1 | 1 | 2
  Argentina | 23 | 20 | 43
  Brazil | 72 | 73 | 145
  Colombia | 10 | 9 | 19
  Venezuela | 4 | 3 | 7
  Mexico | 14 | 15 | 29
  Finland | 1 | 2 | 3
  Germany | 14 | 14 | 28
Origin [Number; unit: participants]
  Caucasian | 153 | 148 | 301
  Non-Caucasian | 61 | 66 | 127
Prior Bisphosphonate User [Number; unit: participants]
  Yes | 20 | 20 | 40
  No | 194 | 194 | 388
Baseline Biochemical Markers of Bone Metabolism [Mean (Standard Deviation); unit: ug/L]
  Serum N-terminal propeptide of type 1 procollagen | 46.161 (35.471) | 47.235 (29.606) | 46.704 (32.562)
  Procollagen I carboxy-terminal propeptide | 166.402 (99.625) | 152.109 (56.637) | 158.845 (79.910)
  Bone-specific alkaline phosphatase | 9.465 (4.522) | 9.711 (4.527) | 9.595 (4.513)
  Osteocalcin | 17.130 (14.422) | 15.878 (10.286) | 16.492 (12.468)
Baseline Bone Mineral Density [Mean (Standard Deviation); unit: grams per square centimeters]
  Lumbar Spine Bone Mineral Density | 0.845 (0.131) | 0.844 (0.128) | 0.845 (0.129)
  Total Hip Bone Mineral Density | 0.744 (0.113) | 0.757 (0.124) | 0.750 (0.119)
  Femoral Neck Bone Mineral Density | 0.682 (0.114) | 0.697 (0.119) | 0.689 (0.116)
C-terminal telopeptide of type I collagen [Mean (Standard Deviation); unit: pmol/L] | 3790.483 (2478.189) | 4543.156 (4838.919) | 4185.328 (3907.204)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at 18 Month Endpoint in Lumbar Spine Bone Mineral Density (BMD)
Description: change from baseline at endpoint in bone mineral density of the lumbar spine as assessed by dual energy X-ray absorptiometry (DXA)
Time Frame: 18 month endpoint
Population: The intention-to-treat analysis was performed using all randomized and treated patients.
Measure: Least Squares Mean (Standard Error); unit: grams per square centimeters
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 198 | 195
grams per square centimeters | 0.059 (0.006) | 0.028 (0.006)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; This is a last observation carried forward analysis that included all patients with a baseline and at least one postbaseline lumbar spine bone mineral density (BMD) measurement; Test type: Superiority or Other; p < 0.001, ANOVA — All comparisons were conducted using a 2-sided significance level of 0.05; ANOVA Model: Change in BMD=treatment+region+prior bisphosponate use+gender. Least Squares Means from treatment

2. Secondary Outcome: Change From Baseline at 18 Month Endpoint in Lumbar Spine Bone Mineral Density (BMD), Female Subset
Description: as for outcome 1
Time Frame: 18 month endpoint
Population: The intention-to-treat analysis was performed using all randomized and treated patients (female only subset).
Measure: Least Squares Mean (Standard Error); unit: grams per square centimeters
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 160 | 159
grams per square centimeters | 0.056 (0.006) | 0.023 (0.006)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — All comparisons were conducted using a 2-sided significance level of 0.05; ANOVA Model: Change in BMD=treatment+region+prior bisphosponate use. Least Squares Means from treatment

3. Secondary Outcome: Time Course of Change From Baseline in Lumbar Spine Bone Mineral Density (BMD), Women and Men Combined
Description: change from baseline in bone mineral density of the lumbar spine as assessed by dual energy X-ray absorptiometry (DXA)
Time Frame: 3, 6, 12, 18, 24, 36 months
Population: The intention-to-treat analysis was performed using all randomized and treated patients. No missing data were imputed.
Measure: Least Squares Mean (Standard Error); unit: grams per square centimeters
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 198 | 195
grams per square centimeters
  Change from baseline at Month 36 (N=123,N=112) | 0.090 (0.006) | 0.044 (0.007)
  Change from baseline at Month 24 (N=136,N=131) | 0.081 (0.006) | 0.043 (0.006)
  Change from baseline at Month 18 (N=156,N=148) | 0.066 (0.005) | 0.031 (0.005)
  Change from baseline at Month 12 (N=170,N=159) | 0.054 (0.004) | 0.028 (0.004)
  Change from baseline at Month 6 (N=178,N=173) | 0.034 (0.004) | 0.018 (0.004)
  Change from baseline at Month 3 (N=183,N=184) | 0.019 (0.004) | 0.012 (0.004)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; Mixed Model Repeated Measures: Change in BMD=treatment+region+prior bisphosphonate use+gender+baseline BMD+visit+treatment*visit; Test type: Superiority or Other; p = 0.058, Mixed Models Analysis — P-value for Month 3; Least Squares Means obtained from the treatment*visit interaction term from the above mixed model repeated measures model
Statistical Analysis 2: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 6 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 12 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 18 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 24 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 36 months; [statistical method as in outcome 3, analysis 1]

4. Secondary Outcome: Time Course of Change From Baseline in Lumbar Spine Bone Mineral Density (BMD), Female Subset
Description: change from baseline in bone mineral density of the lumbar spine as assessed by dual energy X-ray absorptiometry (DXA)
Time Frame: 3, 6, 12, and 18 months
Population: The intention-to-treat analysis was performed using all randomized and treated patients. No missing data were imputed.
Measure: Least Squares Mean (Standard Error); unit: grams per square centimeters
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 172 | 173
grams per square centimeters
  Change from baseline at Month 18 (N=127,N=119) | 0.062 (0.005) | 0.027 (0.005)
  Change from baseline at Month 12 (N=139,N=129) | 0.052 (0.004) | 0.024 (0.004)
  Change from baseline at Month 6 (N=147,N=139) | 0.031 (0.004) | 0.015 (0.004)
  Change from baseline at Month 3 (N=149,N=150) | 0.017 (0.004) | 0.012 (0.004)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.120, Mixed Models Analysis — P-value for 3 Months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 6 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 12 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 18 months; [statistical method as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline in Lumbar Spine Bone Mineral Density (BMD), Women and Men Combined
Description: change from baseline in bone mineral density of the lumbar spine as assessed by dual energy X-ray absorptiometry (DXA)
Time Frame: 24 and 36 months and Endpoint at 36 months
Population: The intention-to-treat analysis was performed using all randomized and treated patients. For 24 and 36 month time points, no missing data were imputed. However, at the 36 month endpoint, last observation carried forward analysis was applied.
Measure: Least Squares Mean (Standard Error); unit: grams per square centimeters
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 198 | 195
grams per square centimeters
  Change, baseline to 36 month endpoint(N=198,N=195) | 0.073 (0.008) | 0.034 (0.008)
  Change from baseline at 36 months (N=123, N=112) | 0.090 (0.006) | 0.044 (0.007)
  Change from baseline at 24 months (N=136, N=131) | 0.081 (0.006) | 0.043 (0.006)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — p-value for 36 month endpoint; ANOVA Model: Change in BMD=treatment+region+prior bisphosponate use+gender. Least Squares Means from treatment
Statistical Analysis 2: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — p-value for 36 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 24 months; [statistical method as in outcome 3, analysis 1]

6. Secondary Outcome: Change From Baseline in Femoral Neck Bone Mineral Density (BMD), Women and Men Combined
Description: change from baseline in bone mineral density of the femoral neck as assessed by dual energy X-ray absorptiometry (DXA)
Time Frame: 18, 24, 36 months, and 18 and 36 month endpoints
Population: The intention-to-treat analysis was performed using all randomized and treated patients. For 18, 24 and 36 month time points, no missing data were imputed. However at the 36 month endpoint, last observation carried forward analysis was applied.
Measure: Least Squares Mean (Standard Error); unit: grams per square centimeters
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 185 | 177
grams per square centimeters
  Change, baseline to 36 month endpoint(N=185,N=177) | 0.033 (0.006) | 0.017 (0.006)
  Change from baseline at 36 months(N=120,N=113) | 0.041 (0.005) | 0.021 (0.005)
  Change from baseline at 24 months(N=135,N=131) | 0.030 (0.005) | 0.015 (0.005)
  Change, baseline to 18 month endpoint(N=185,N=176) | 0.024 (0.005) | 0.014 (0.005)
  Change from baseline at 18 months (N=156,N=145) | 0.028 (0.005) | 0.017 (0.005)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; This is a last observation carried forward analysis that included all patients with a baseline and at least one postbaseline femoral neck bone mineral density (BMD) measurement; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for 36-month endpoint; ANOVA Model: Change in BMD=treatment+region+prior bisphosponate use+gender. Least Squares Means from treatment
Statistical Analysis 2: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 36 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — P-value for 24 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.011, ANOVA — P-value for 18 month endpoint; ANOVA Model: Change in BMD=treatment+region+prior bisphosponate use+gender. Least Squares Means from treatment
Statistical Analysis 5: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis — P-value for 18 months; [statistical method as in outcome 3, analysis 1]

7. Secondary Outcome: Change From Baseline in Total Hip Bone Mineral Density (BMD), Women and Men Combined
Description: change from baseline in bone mineral density of the total hip as assessed by dual energy X-ray absorptiometry (DXA)
Time Frame: 18, 24, 36 months, and 18 and 36 month endpoints
Population: The intention-to-treat analysis was performed using all randomized and treated patients. For 18, 24 and 36 month time points, no missing data were imputed. However, at 18 and 36 month endpoints, last observation carried forward analyses were applied.
Measure: Least Squares Mean (Standard Error); unit: grams per square centimeters
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 185 | 177
grams per square centimeters
  Change, baseline to 36 month endpoint(N=185,N=177) | 0.032 (0.005) | 0.017 (0.005)
  Change from baseline at 36 months(N=120,N=113) | 0.037 (0.005) | 0.020 (0.005)
  Change from baseline at 24 months(N=135,N=131) | 0.034 (0.004) | 0.018 (0.004)
  Change, baseline to 18 month endpoint(N=185,N=176) | 0.026 (0.004) | 0.017 (0.004)
  Change from baseline at 18 months (N=156,N=144) | 0.027 (0.004) | 0.018 (0.004)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; This is a last observation carried forward analysis that included all patients with a baseline and at least one postbaseline total hip bone mineral density (BMD) measurement; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for 36 month endpoint; ANOVA Model: Change in BMD=treatment+region+prior bisphosponate use+gender. Least Squares Means from treatment
Statistical Analysis 2: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 36 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 24 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.006, ANOVA — P-value for 18 month endpoint; ANOVA Model: Change in BMD=treatment+region+prior bisphosponate use+gender. Least Squares Means from treatment
Statistical Analysis 5: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis — P-value for 18 months; [statistical method as in outcome 3, analysis 1]

8. Secondary Outcome: Time Course of Change From Baseline in Femoral Neck Bone Mineral Density (BMD), Women and Men Combined
Description: change from baseline in bone mineral density of the femoral neck as assessed by dual energy X-ray absorptiometry (DXA)
Time Frame: 12, 18, 24, and 36 months
Population: The intention-to-treat analysis was performed using all randomized and treated patients. No missing data were imputed.
Measure: Least Squares Mean (Standard Error); unit: grams per square centimeters
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 185 | 177
grams per square centimeters
  Change from baseline at Month 36 (N=120,N=113) | 0.041 (0.005) | 0.021 (0.005)
  Change from baseline at Month 24 (N=135,N=131) | 0.030 (0.005) | 0.015 (0.005)
  Change from baseline at Month 18 (N=156,N=145) | 0.028 (0.005) | 0.017 (0.005)
  Change from baseline at Month 12 (N=167,N=158) | 0.026 (0.005) | 0.012 (0.005)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 12 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis — P-value for 18 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — P-value for 24 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 36 months; [statistical method as in outcome 3, analysis 1]

9. Secondary Outcome: Time Course of Change From Baseline in Total Hip Bone Mineral Density (BMD), Women and Men Combined
Description: change from baseline in bone mineral density of the total hip as assessed by dual energy X-ray absorptiometry (DXA)
Time Frame: 12, 18, 24, and 36 months
Population: The intention-to-treat analysis was performed using all randomized and treated patients. No missing data was imputed.
Measure: Least Squares Mean (Standard Error); unit: grams per square centimeters
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 185 | 177
grams per square centimeters
  Change from baseline at 36 Months (N=120, N=113) | 0.037 (0.005) | 0.020 (0.005)
  Change from baseline at 24 Months (N=135, N=131) | 0.034 (0.004) | 0.018 (0.004)
  Change from baseline at 18 Months (N=156, N=145) | 0.027 (0.004) | 0.018 (0.004)
  Change from baseline at 12 Months (N=167, N=158) | 0.022 (0.004) | 0.014 (0.004)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — P-value for 12 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis — P-value for 18 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 24 months; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Teriparatide vs Alendronate; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for 36 months; [statistical method as in outcome 3, analysis 1]

10. Secondary Outcome: Time Course of Change From Baseline in Bone Turnover Markers in Subset of Patients - Serum N-terminal Propeptide of Type 1 Procollagen
Time Frame: 1, 6, 18, and 36 months
Population: Subset of patients with measures of biochemical markers
Measure: Mean (Standard Error); unit: percent
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 99 | 100
percent
  Percent change from baseline at Month 1(N=98,N=99) | 107.0 (13.744) | -14.8 (2.861)
  Percent change from baseline at Month 6(N=86,N=85) | 130.8 (20.752) | -43.2 (3.481)
  Percent change from baseline at Month18(N=77,N=76) | 86.3 (20.231) | -35.8 (4.477)
  Percent change from baseline at Month36(N=59,N=57) | 61.7 (16.156) | -20.2 (10.587)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 1; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 2: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 6; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 3: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 18; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 4: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 36; Wilcoxon Rank Sum Test using the aligned ranks for scores

11. Secondary Outcome: Time Course of Change From Baseline in Bone Turnover Markers in Subset of Patients - Serum C-terminal Propeptide of Type 1 Procollagen
Time Frame: 1, 6, 18, and 36 months
Population: Subset of patients with measures of biochemical markers.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 78 | 89
percent
  Percent change from baseline at Month 1(N=66,N=78) | 48.2 (7.024) | -8.8 (2.912)
  Percent change from baseline at Month 6(N=67,N=76) | 10.5 (5.318) | -22.3 (3.694)
  Percent change from baseline at Month18(N=55,N=65) | 5.1 (8.604) | -21.3 (4.207)
  Percent change from baseline at Month36(N=45,N=49) | -1.3 (7.082) | -15.4 (7.394)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 1; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 2: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 6; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 3: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney) — P-value for Month 18; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 4: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p = 0.013, Wilcoxon (Mann-Whitney) — P-value for Month 36; Wilcoxon Rank Sum Test using the aligned ranks for scores

12. Secondary Outcome: Time Course of Change From Baseline in Bone Turnover Markers in Subset of Patients - Bone-Specific Alkaline Phosphatase
Time Frame: 1, 6, 18, and 36 months
Population: Subset of patients with measures of biochemical markers
Measure: Mean (Standard Error); unit: percent
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 77 | 89
percent
  Percent change from baseline at Month 1(N=65,N=78) | 35.0 (7.518) | 0.5 (4.897)
  Percent change from baseline at Month 6(N=66,N=76) | 52.3 (10.995) | -7.2 (12.384)
  Percent change from baseline at Month18(N=54,N=65) | 34.4 (9.548) | -4.1 (10.501)
  Percent change from baseline at Month36(N=44,N=49) | 44.7 (14.357) | 20.6 (19.912)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 1; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 2: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 6; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 3: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 18; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 4: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 36; Wilcoxon Rank Sum Test using the aligned ranks for scores

13. Secondary Outcome: Time Course of Change From Baseline in Bone Turnover Markers in Subset of Patients - Serum Type 1 Collagen Degradation Fragments
Time Frame: 1, 6, 18, and 36 months
Population: Subset of patients with measures of biochemical markers
Measure: Mean (Standard Error); unit: percent
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 84 | 91
percent
  Percent change from baseline at Month 1(N=70,N=79) | 29.0 (8.192) | -38.6 (4.110)
  Percent change from baseline at Month 6(N=66,N=75) | 66.8 (17.143) | -42.4 (5.050)
  Percent change from baseline at Month18(N=64,N=71) | 29.1 (11.714) | -47.5 (6.305)
  Percent change from baseline at Month36(N=49,N=48) | 30.7 (14.205) | -16.2 (23.178)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 1; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 2: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 6; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 3: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 18; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 4: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 36; Wilcoxon Rank Sum Test using the aligned ranks for scores

14. Secondary Outcome: Time Course of Change From Baseline in Bone Turnover Markers in Subset of Patients - Osteocalcin
Time Frame: 1, 6, 18, and 36 months
Population: Subset of patients with measures of biochemical markers
Measure: Mean (Standard Error); unit: percent
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 97 | 101
percent
  Percent change from baseline at Month1(N=94,N=100) | 147.1 (26.408) | -5.2 (3.447)
  Percent change from baseline at Month 6(N=84,N=88) | 120.0 (16.713) | -33.6 (3.656)
  Percent change from baseline at Month18(N=77,N=77) | 108.9 (22.750) | -25.0 (5.118)
  Percent change from baseline at Month36(N=56,N=58) | 62.1 (20.929) | -19.6 (12.980)
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value for Month 1; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 2: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value at Month 6; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 3: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value at Month 18; Wilcoxon Rank Sum Test using the aligned ranks for scores
Statistical Analysis 4: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value at Month 36; Wilcoxon Rank Sum Test using the aligned ranks for scores

15. Secondary Outcome: Any Fracture, Nonvertebral Fractures, Vertebral Fractures, Clinical Vertebral Fractures, and Severity Fractures
Description: Clinical vertebral fracture was defined as a radiographically confirmed fracture that was associated with symptoms such as back pain.
Time Frame: 36 months
Population: For vertebral fractures, only those patients with baseline and postbaseline spinal radiographs were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Teriparatide | Alendronate
Number analyzed (Participants) | 214 | 214
participants
  Any Fracture | 19 | 27
  Nonvertebral Fracture | 16 | 15
  Vertebral Fracture | 3 | 13
  Clinical Vertebral Fracture | 0 | 4
  Nonvertebral Fragility Fracture | 9 | 5
  Severity-Radiographic Vertebral Fracture: Mild | 1 | 7
  Severity-Radiographic Vertebral Fracture: Moderate | 2 | 2
  Severity-Radiographic Vertebral Fracture: Severe | 0 | 4
Statistical Analysis 1: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p = 0.212, Cochran-Mantel-Haenszel — p-value for Any Fracture
Statistical Analysis 2: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p = 0.843, Cochran-Mantel-Haenszel — p-value for Nonvertebral Fracture
Statistical Analysis 3: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel — p-value for Vertebral Fracture
Statistical Analysis 4: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p = 0.037, Cochran-Mantel-Haenszel — p-value for Clinical Vertebral Fracture
Statistical Analysis 5: Comparison: Teriparatide vs Alendronate; Test type: Superiority or Other; p = 0.256, Cochran-Mantel-Haenszel — p-value for Nonvertebral Fragility Fracture

ADVERSE EVENTS:
Arm/Group | Teriparatide | Alendronate
Serious Adverse Events (participants affected / at risk) | 70 | 64
Other Adverse Events (participants affected / at risk) | 190 | 177
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Teriparatide | Alendronate
Anaemia (Blood and lymphatic system disorders) | 2/214 (2) | 1/214 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0/214 (0) | 1/214 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1/214 (1) | 0/214 (0)
Acute myocardial infarction (Cardiac disorders) | 1/214 (1) | 0/214 (0)
Angina pectoris (Cardiac disorders) | 1/214 (3) | 1/214 (1)
Atrial fibrillation (Cardiac disorders) | 1/214 (1) | 0/214 (0)
Cardiac arrest (Cardiac disorders) | 1/214 (1) | 0/214 (0)
Cardiac failure (Cardiac disorders) | 0/214 (0) | 1/214 (1)
Cardiac failure congestive (Cardiac disorders) | 0/214 (0) | 2/214 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0/214 (0) | 1/214 (1)
Coronary artery disease (Cardiac disorders) | 0/214 (0) | 1/214 (1)
Myocardial infarction (Cardiac disorders) | 2/214 (2) | 2/214 (2)
Ventricular fibrillation (Cardiac disorders) | 1/214 (1) | 0/214 (0)
Epidermolysis (Congenital, familial and genetic disorders) | 1/214 (1) | 0/214 (0)
Adrenal insufficiency (Endocrine disorders) | 1/214 (1) | 0/214 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0/214 (0) | 1/214 (1)
Blindness (Eye disorders) | 1/214 (1) | 0/214 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1/214 (1) | 0/214 (0)
Abdominal pain (Gastrointestinal disorders) | 0/214 (0) | 1/214 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0/214 (0) | 1/214 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0/214 (0) | 1/214 (2)
Colitis ulcerative (Gastrointestinal disorders) | 1/214 (1) | 0/214 (0)
Constipation (Gastrointestinal disorders) | 2/214 (2) | 0/214 (0)
Diarrhoea (Gastrointestinal disorders) | 0/214 (0) | 1/214 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1/214 (1) | 0/214 (0)
Gastric ulcer (Gastrointestinal disorders) | 0/214 (0) | 1/214 (1)
Gastritis (Gastrointestinal disorders) | 2/214 (2) | 0/214 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/214 (1) | 1/214 (1)
Hiatus hernia (Gastrointestinal disorders) | 0/214 (0) | 1/214 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/214 (0) | 1/214 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 0/214 (0) | 1/214 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1/214 (1) | 0/214 (0)
Subileus (Gastrointestinal disorders) | 1/214 (1) | 0/214 (0)
Vomiting (Gastrointestinal disorders) | 0/214 (0) | 1/214 (1)
Asthenia (General disorders) | 0/214 (0) | 1/214 (1)
Chest pain (General disorders) | 1/214 (1) | 0/214 (0)
Death (General disorders) | 2/214 (2) | 4/214 (4)
Impaired healing (General disorders) | 1/214 (1) | 0/214 (0)
Multi-organ failure (General disorders) | 0/214 (0) | 1/214 (1)
Pain (General disorders) | 0/214 (0) | 1/214 (1)
Ulcer (General disorders) | 1/214 (1) | 0/214 (0)
Cholecystitis (Hepatobiliary disorders) | 1/214 (1) | 0/214 (0)
Cholelithiasis (Hepatobiliary disorders) | 1/214 (1) | 1/214 (1)
Antiphospholipid syndrome (Immune system disorders) | 0/214 (0) | 1/214 (1)
Sarcoidosis (Immune system disorders) | 1/214 (1) | 0/214 (0)
Abscess (Infections and infestations) | 0/214 (0) | 1/214 (1)
Abscess bacterial (Infections and infestations) | 0/214 (0) | 1/214 (1)
Arthritis bacterial (Infections and infestations) | 1/214 (1) | 1/214 (1)
Bronchitis (Infections and infestations) | 0/214 (0) | 1/214 (1)
Bronchopneumonia (Infections and infestations) | 0/214 (0) | 2/214 (6)
Cardiac infection (Infections and infestations) | 0/214 (0) | 1/214 (1)
Cellulitis (Infections and infestations) | 3/214 (3) | 3/214 (3)
Chronic sinusitis (Infections and infestations) | 1/214 (1) | 0/214 (0)
Corneal infection (Infections and infestations) | 1/214 (1) | 0/214 (0)
Escherichia infection (Infections and infestations) | 1/214 (1) | 0/214 (0)
Gastroenteritis (Infections and infestations) | 0/214 (0) | 2/214 (2)
Gastroenteritis salmonella (Infections and infestations) | 1/214 (1) | 0/214 (0)
Gastrointestinal infection (Infections and infestations) | 1/214 (1) | 0/214 (0)
Herpes zoster (Infections and infestations) | 2/214 (2) | 0/214 (0)
Intervertebral discitis (Infections and infestations) | 1/214 (1) | 0/214 (0)
Labyrinthitis (Infections and infestations) | 0/214 (0) | 1/214 (1)
Lobar pneumonia (Infections and infestations) | 2/214 (2) | 1/214 (1)
Lung abscess (Infections and infestations) | 1/214 (1) | 0/214 (0)
Lung infection (Infections and infestations) | 0/214 (0) | 1/214 (1)
Osteomyelitis (Infections and infestations) | 1/214 (1) | 0/214 (0)
Pneumonia (Infections and infestations) | 8/214 (8) | 6/214 (6)
Pneumonia staphylococcal (Infections and infestations) | 1/214 (1) | 0/214 (0)
Pneumonia streptococcal (Infections and infestations) | 1/214 (1) | 0/214 (0)
Pulmonary tuberculosis (Infections and infestations) | 1/214 (1) | 0/214 (0)
Respiratory tract infection (Infections and infestations) | 1/214 (1) | 0/214 (0)
Salmonella sepsis (Infections and infestations) | 1/214 (1) | 0/214 (0)
Sepsis (Infections and infestations) | 2/214 (2) | 2/214 (2)
Septic shock (Infections and infestations) | 2/214 (2) | 2/214 (2)
Sinusitis (Infections and infestations) | 0/214 (0) | 1/214 (1)
Tracheobronchitis (Infections and infestations) | 0/214 (0) | 1/214 (1)
Urinary tract infection (Infections and infestations) | 2/214 (2) | 4/214 (5)
Urosepsis (Infections and infestations) | 0/214 (0) | 1/214 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0/214 (0) | 1/214 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0/214 (0) | 1/214 (1)
Device failure (Injury, poisoning and procedural complications) | 0/214 (0) | 1/214 (1)
Fall (Injury, poisoning and procedural complications) | 3/214 (3) | 3/214 (3)
Forearm fracture (Injury, poisoning and procedural complications) | 1/214 (1) | 0/214 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0/214 (0) | 1/214 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0/214 (0) | 1/214 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0/214 (0) | 1/214 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1/214 (1) | 0/214 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1/214 (1) | 1/214 (1)
Renal injury (Injury, poisoning and procedural complications) | 1/214 (1) | 0/214 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1/214 (1) | 0/214 (0)
Suture rupture (Injury, poisoning and procedural complications) | 1/214 (1) | 0/214 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0/214 (0) | 1/214 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1/214 (1) | 0/214 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0/214 (0) | 1/214 (1)
Dehydration (Metabolism and nutrition disorders) | 0/214 (0) | 1/214 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0/214 (0) | 1/214 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0/214 (0) | 1/214 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1/214 (2) | 0/214 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2/214 (3) | 0/214 (0)
Obesity (Metabolism and nutrition disorders) | 1/214 (1) | 0/214 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/214 (1) | 1/214 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1/214 (1) | 0/214 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0/214 (0) | 1/214 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0/214 (0) | 1/214 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0/214 (0) | 1/214 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3/214 (3) | 2/214 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1/214 (1) | 0/214 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/214 (1) | 0/214 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1/214 (1) | 0/214 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/214 (0) | 1/214 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/214 (1) | 0/214 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/214 (0) | 1/214 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/214 (1) | 0/214 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/214 (1) | 0/214 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/214 (0) | 1/214 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/214 (0) | 1/214 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/214 (1) | 0/214 (0)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/214 (0) | 1/214 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/214 (1) | 0/214 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/214 (1) | 0/214 (0)
Cerebrovascular accident (Nervous system disorders) | 0/214 (0) | 1/214 (1)
Cervical myelopathy (Nervous system disorders) | 0/214 (0) | 1/214 (1)
Headache (Nervous system disorders) | 1/214 (1) | 0/214 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0/214 (0) | 1/214 (1)
Paraesthesia (Nervous system disorders) | 1/214 (1) | 0/214 (0)
Sensory disturbance (Nervous system disorders) | 1/214 (1) | 0/214 (0)
Syncope (Nervous system disorders) | 1/214 (1) | 1/214 (1)
Transient ischaemic attack (Nervous system disorders) | 0/214 (0) | 1/214 (1)
Agitation (Psychiatric disorders) | 0/214 (0) | 1/214 (1)
Confusional state (Psychiatric disorders) | 1/214 (1) | 0/214 (0)
Delusion (Psychiatric disorders) | 0/214 (0) | 1/214 (1)
Depression (Psychiatric disorders) | 1/214 (1) | 0/214 (0)
Haematuria (Renal and urinary disorders) | 0/214 (0) | 1/214 (1)
Hydronephrosis (Renal and urinary disorders) | 1/214 (1) | 0/214 (0)
Nephrolithiasis (Renal and urinary disorders) | 1/214 (1) | 0/214 (0)
Renal failure acute (Renal and urinary disorders) | 2/214 (2) | 1/214 (1)
Renal failure chronic (Renal and urinary disorders) | 1/214 (1) | 0/214 (0)
Ureteric obstruction (Renal and urinary disorders) | 1/214 (1) | 0/214 (0)
Prostatic intraepithelial neoplasia (Reproductive system and breast disorders) | 1/214 (1) | 0/214 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/214 (1) | 0/214 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/214 (1) | 0/214 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5/214 (9) | 2/214 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4/214 (4) | 2/214 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0/214 (0) | 1/214 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0/214 (0) | 1/214 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0/214 (0) | 1/214 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1/214 (1) | 0/214 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1/214 (1) | 0/214 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1/214 (1) | 0/214 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3/214 (3) | 2/214 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1/214 (1) | 1/214 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0/214 (0) | 2/214 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2/214 (2) | 2/214 (2)
Panniculitis (Skin and subcutaneous tissue disorders) | 1/214 (1) | 0/214 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0/214 (0) | 1/214 (1)
Arthrodesis (Surgical and medical procedures) | 0/214 (0) | 1/214 (1)
Coronary artery bypass (Surgical and medical procedures) | 1/214 (1) | 0/214 (0)
Hip arthroplasty (Surgical and medical procedures) | 3/214 (3) | 0/214 (0)
Knee arthroplasty (Surgical and medical procedures) | 3/214 (4) | 1/214 (2)
Surgery (Surgical and medical procedures) | 1/214 (1) | 0/214 (0)
Thyroidectomy (Surgical and medical procedures) | 0/214 (0) | 1/214 (1)
Vertebroplasty (Surgical and medical procedures) | 0/214 (0) | 2/214 (2)
Arterial insufficiency (Vascular disorders) | 0/214 (0) | 1/214 (1)
Arterial occlusive disease (Vascular disorders) | 1/214 (1) | 0/214 (0)
Deep vein thrombosis (Vascular disorders) | 2/214 (2) | 1/214 (1)
Haematoma (Vascular disorders) | 1/214 (1) | 0/214 (0)
Hypertension (Vascular disorders) | 0/214 (0) | 1/214 (1)
Peripheral vascular disorder (Vascular disorders) | 1/214 (1) | 0/214 (0)
Shock (Vascular disorders) | 0/214 (0) | 1/214 (1)
Thrombophlebitis (Vascular disorders) | 0/214 (0) | 1/214 (1)
Venous thrombosis (Vascular disorders) | 1/214 (1) | 0/214 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Teriparatide | Alendronate
Anaemia (Blood and lymphatic system disorders) | 10/214 (10) | 16/214 (16)
Abdominal pain (Gastrointestinal disorders) | 11/214 (12) | 10/214 (12)
Abdominal pain upper (Gastrointestinal disorders) | 18/214 (19) | 16/214 (16)
Dyspepsia (Gastrointestinal disorders) | 9/214 (9) | 15/214 (16)
Gastritis (Gastrointestinal disorders) | 15/214 (15) | 8/214 (8)
Nausea (Gastrointestinal disorders) | 36/214 (44) | 18/214 (23)
Vomiting (Gastrointestinal disorders) | 13/214 (13) | 11/214 (12)
Bronchitis (Infections and infestations) | 20/214 (32) | 17/214 (22)
Influenza (Infections and infestations) | 18/214 (24) | 24/214 (29)
Nasopharyngitis (Infections and infestations) | 7/214 (8) | 13/214 (21)
Sinusitis (Infections and infestations) | 15/214 (23) | 18/214 (24)
Urinary tract infection (Infections and infestations) | 20/214 (27) | 26/214 (31)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21/214 (26) | 19/214 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 24/214 (25) | 26/214 (28)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10/214 (12) | 12/214 (15)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 15/214 (15) | 18/214 (18)
Dizziness (Nervous system disorders) | 17/214 (20) | 15/214 (15)
Headache (Nervous system disorders) | 18/214 (23) | 14/214 (17)
Depression (Psychiatric disorders) | 18/214 (19) | 16/214 (16)
Insomnia (Psychiatric disorders) | 12/214 (12) | 3/214 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13/214 (17) | 4/214 (6)
Hypertension (Vascular disorders) | 21/214 (21) | 18/214 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days